CLINICAL TRIAL: NCT03906968
Title: SinuSonic Study for Adults With Nasal Congestion
Brief Title: The Safety and Efficacy of a SinuSonic Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00083883
Record Dates: First submitted 2019-03-26; First posted 2019-04-08 (Actual); Results first posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Nasal Congestion
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- SinuSonic Device (Experimental): SinuSonic Device used twice a day for four to six weeks.
  Interventions: Device: SinuSonic Device

INTERVENTIONS:
Device: SinuSonic Device — A medical device that utilizes sound and pressure combined with normal breathing to relieve nasal congestion

SUMMARY:
This study aims to test the safety and effectiveness of the SinuSonic device on adults with moderate to severe nasal congestion. SinuSonic is a medical device that utilizes sound and pressure combined with normal breathing to relieve nasal congestion. This device is held over the nose for 3 minutes. This study will use patient responses to measure how effective SinuSonic devices are in treating these moderate to severe congestion in adults. The study will consist of 40 subjects at the Medical University of South Carolina and will take place over the course of 4 to 6 weeks starting with a baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age
2. Complaints of nasal congestion present for 2 weeks or more and a qualifying nasal congestion score of >5 (10 point VAS scale)

Exclusion Criteria:

1. Fixed structural cause of nasal congestion (moderate or severe septal deviation, moderate or severe nasal valve collapse, Grade 3-4 polyp)
2. Inability to read and understand English
3. Allergic sensitivity to silicone or any other component of device
4. History of severe nose bleeding within last 3 months
5. Anticoagulation (Aspirin is acceptable)
6. Known pregnancy
7. Current nasal crusting or ulceration revealed on rhinoscopy
8. Inability to perform treatment due to underlying medical condition
9. Topical decongestant use in last week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-31 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary M Soler, Principal Investigator — Medical University of South Carolina
Locations (1):
- Sinus Center - Medical Univesity of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Not Applicable. We plan to publish this study.

REFERENCES:
- [Derived] Soler ZM, Nguyen SA, Salvador C, Lackland T, Desiato VM, Storck K, Schlosser RJ. A novel device combining acoustic vibration with oscillating expiratory pressure for the treatment of nasal congestion. Int Forum Allergy Rhinol. 2020 May;10(5):610-618. doi: 10.1002/alr.22537. Epub 2020 Feb 27. PMID 32104962

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SinuSonic Device
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SinuSonic Device
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants] — > 18 years old
  Participants
    <=18 years | 0
    Between 18 and 65 years | 39
    >=65 years | 1
Age, Continuous [Mean (Full Range); unit: Years] | 39.1 [20 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 26
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 40
visual analogue scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — The visual analog scale (VAS) for rhinosinusitis is used to evaluate the total severity. The subject is asked to indicate on a VAS the answer to the question: "How troublesome are your symptoms of rhinosinusitis?" Subject will assess Nasal symptoms using a 10 cm Visual Analog Scale for each symptom, 0=not troublesome and 10 = the worst imaginable. The disease can be divided into Mild, Moderate and Severe based on total severity VAS score (0 to 10 cm):
  Mild = VAS 0-3 Moderate = VAS > 3-7 Severe = VAS > 7-10
  units on a scale | 5.8 (2.4)
Total Nasal Symptom Score (TNSS) [Mean (Standard Deviation); unit: units on a scale] — Change from baseline to week 6 in subject congestion symptom severity, as measured by the Total Nasal Symptom Score (TNSS, range 0-3). Where 0 indicates no symptoms, a score of 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity. TNSS is calculated by adding the score for each of the symptoms to a total out of 15.
  units on a scale | 7.2 (3.5)
Nasal Obstruction and Septoplasty Effectiveness (NOSE) score [Mean (Standard Deviation); unit: units on a scale] — Change from baseline to week 6 in subject nasal congestion severity, as measured by the Nasal Obstruction and Septoplasty Effectiveness Scale (NOSE Scale). The NOSE scale is a subject-completed questionnaire that consists of 5 questions. Each item is rated as follows: 0=not a problem, 1=very mild problem, 2=moderate problem, 3=fairly bad problem, 4=severe problem. The total score can range from 0-100, 0 being the best and 100 being the worst.
  units on a scale | 50.4 (19.9)
22-item Sino-Nasal Outcome Test (SNOT-22) [Mean (Standard Deviation); unit: units on a scale] — Change from baseline to week 6 in subject symptoms and functioning, as measured by Sinonasal Outcome Test - 22 (SNOT-22). SNOT-22 is a subject-completed questionnaire that consists of 22 questions. Each item is rated as follows: 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be. The total score can range from 0-110, 0 being the best and 110 being the worst.
  units on a scale | 31.7 (20.3)
peak nasal inspiratory flow (PNIF) [Median (Standard Deviation); unit: L/min] | 79.5 (43.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Nasal Symptom Score (TNSS) at 4 to 6 Weeks
Description: Change from baseline to week 6 in subject congestion symptom severity, as measured by the Total Nasal Symptom Score (TNSS, range 0-3). Where 0 indicates no symptoms, a score of 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity. TNSS is calculated by adding the score for each of the symptoms to a total out of 15.
Time Frame: Total Nasal Symptom Score (TNSS) at 4 to 6 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SinuSonic Device
Number analyzed (Participants) | 40
score on a scale | 3.5 (3.1)

2. Secondary Outcome: Change in Peak Nasal Inspiratory Flow Test (PNIF Test)
Description: Change from baseline to week 2 in subject nasal airway obstruction, as measure by the Peak Nasal Inspiratory Flow Test (PNIF Test). The PNIF is used to diagnose the patency of the nose.
Time Frame: Peak Nasal Inspiratory Flow Test (PNIF Test) score at 2 Weeks
Measure: Median (Standard Deviation); unit: L/min
Arm/Group | SinuSonic Device
Number analyzed (Participants) | 40
L/min | 104.5 (41.3)

3. Secondary Outcome: Change in Sinonasal Outcome Test 22 (SNOT-22) Total Score
Description: Change from baseline to week 6 in subject symptoms and functioning, as measured by Sinonasal Outcome Test - 22 (SNOT-22). SNOT-22 is a subject-completed questionnaire that consists of 22 questions. Each item is rated as follows: 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be. The total score can range from 0-110, 0 being the best and 110 being the worst.
Time Frame: Sinonasal Outcome Test 22 (SNOT-22) Total Score at 4 to 6 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SinuSonic Device
Number analyzed (Participants) | 40
score on a scale | 14.2 (12.7)

4. Secondary Outcome: Change in Visual Analog Scale (VAS)
Description: The visual analog scale (VAS) for rhinosinusitis is used to evaluate the total severity. The subject is asked to indicate on a VAS the answer to the question: "How troublesome are your symptoms of rhinosinusitis?" Subject will assess Nasal symptoms using a 10 cm Visual Analog Scale for each symptom, 0=not troublesome and 10 = the worst imaginable. The disease can be divided into Mild, Moderate and Severe based on total severity VAS score (0 to 10 cm):
  * Mild = VAS 0-3
  * Moderate = VAS > 3-7
  * Severe = VAS > 7-10
Time Frame: Visual Analog Scale (VAS) score at 4 to 6 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SinuSonic Device
Number analyzed (Participants) | 40
score on a scale | 2.6 (2.3)

5. Secondary Outcome: Change in Nasal Obstruction and Septoplasty Effectiveness Scale (NOSE Scale)
Description: Change from baseline to week 6 in subject nasal congestion severity, as measured by the Nasal Obstruction and Septoplasty Effectiveness Scale (NOSE Scale). The NOSE scale is a subject-completed questionnaire that consists of 5 questions. Each item is rated as follows: 0=not a problem, 1=very mild problem, 2=moderate problem, 3=fairly bad problem, 4=severe problem. The total score can range from 0-100, 0 being the best and 100 being the worst.
Time Frame: Nasal Obstruction and Septoplasty Effectiveness Scale (NOSE Scale) score at 4 to 6 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SinuSonic Device
Number analyzed (Participants) | 40
score on a scale | 23.3 (17.2)

6. Other Pre Specified Outcome: Safety Descriptive About Occurrence of Adverse Events
Description: Safety will be evaluated by the Adverse events occurence
Time Frame: 4 to 6 Weeks
Measure: Number; unit: reported adverse events
Arm/Group | SinuSonic Device
Number analyzed (Participants) | 40
reported adverse events | 0

7. Other Pre Specified Outcome: Evaluation of Results of General Physical Examination
Description: Collection of safety data throughout the whole study period
Time Frame: 4 to 6 Weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 9 months
Description: This is a minimal risk study based on a commercially available device.
Arm/Group | SinuSonic Device
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT03906968/Prot_SAP_002.pdf
  • Informed Consent Form (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT03906968/ICF_001.pdf